CLINICAL TRIAL: NCT05999981
Title: Comparison Between Ultrasound Guided Transversalis Fascia Plane Block and Transversus Abdominis Plane Block on Postoperative Recovery in Patients Undergoing Cesarean Section Surgery
Brief Title: Comparison of the Quality of Recovery After Cesarean Section Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Melike Korkmaz Toker, Associate Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSKU 13-IV
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Recovery; Abdominal Pain; Cesarean Section
Keywords: cesarean section surgery; postoperative recovery; postoperative pain; trasversalis fascia plane block; transversus abdominis plane block; obstetric quality of recovery 11 Turkish score; numeric rating scale
MeSH Terms: conditions — Abdominal Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversalis Fascia Plane Block (TFPB) Group (Active Comparator): At TFPB group, the block will be performed by ultrasound guidance after completion of surgery. TFPB will be performed under ultrasonography guidance using a linear 6 to 13 megahertz ultrasound probe by the anesthesiologist. In TFPB group patients will receive 40 ml %0.25 bupivacaine divided into 2 equal doses between transversus abdominis muscle and transversalis fascia bilaterally.
  Interventions: Procedure: Transversalis Fascia Plane Block
- Transversus Abdominis Plane (TAP) Block Group (Active Comparator): At TAP block group, the block will be performed by ultrasound guidance after completion of surgery. TAP blocks will be performed under ultrasonography guidance using a linear 6 to 13 megahertz ultrasound probe by the anesthesiologist. In TAP block group patients will receive 40 ml %0.25 bupivacaine divided into 2 equal doses in the fascial plane between internal oblique muscle and transversus abdominis muscle bilaterally.
  Interventions: Procedure: Transversus Abdominis Plane Block

INTERVENTIONS:
Procedure: Transversalis Fascia Plane Block — 40 ml %0.25 bupivacaine divided into 2 equal doses will be injected by the anesthesiologist under ultrasonography guidance between transversus abdominis muscle and transversalis fascia bilaterally
  Arms: Transversalis Fascia Plane Block (TFPB) Group
Procedure: Transversus Abdominis Plane Block — 40 ml %0.25 bupivacaine divided into 2 equal doses will be injected by the anesthesiologist under ultrasonography guidance in the fascial plane between internal oblique muscle and transversus abdominis muscle bilaterally
  Arms: Transversus Abdominis Plane (TAP) Block Group

SUMMARY:
Inadequate pain control after cesarean section surgery causes postpartum depression, persistent pain and delayed mother-infant bonding. The investigator's aim is to asses whether ultrasound guided transversalis fascia plane block (TFPB) or transversus abdominis plane (TAP) block would improve postoperative quality of recovery and decrease postoperative opioid consumption after cesarean section surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status II-III
* Cesarean section surgery under spinal anesthesia

Exclusion Criteria:

* American Society of Anesthesiologists physical status IV
* Emergency surgery
* General anesthesia
* Additional surgical intervention at the same session
* Body mass index of more than 35 kg/m2
* Allergy to any study drugs
* Local infection at the injection site
* History of drug abuse
* Communication problem
* Coagulopathy
* Preeclampsia and eclampsia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Postoperative quality of recovery | Postoperative 24th hour
  Postoperative quality of recovery will be assessed by Obstetric Quality of Recovery 11 Turkish (ObsQoR-11T) score

SECONDARY OUTCOMES:
Postoperative opioid consumption | Postoperative 1st, 2nd, 4th, 8th 12th and 24th hour
  Morphine consumption will be assessed by checking patient controlled analgesia (PCA) device records and fentanyl consumption will be assessed by checking patient daily drug order records
Numeric Rating Scale | Postoperative 1st, 2nd, 4th, 8th 12th and 24th hour
  A blinded nurse will assess postoperative pain during resting and movement at postoperative 1st, 2nd, 4th, 8th 12th and 24th hour by using 11-point Numerical Rating Scale which ranges from '0' (means no pain) to '10' (means worst pain imaginable)
Adverse Reactions | Postoperative 24th hour
  Nausea, vomiting, constipation, urinary retention and skin rash/pruritus will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Melike Korkmaz Toker, Associate Professor, Principal Investigator — Mugla Sıtkı Kocman University Department of Anesthesiology and Reanimation
Locations (1):
- Mugla Sıtkı Kocman University Training and Research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
via mail

REFERENCES:
- [Background] Jadon A, Jain P, Chakraborty S, Motaka M, Parida SS, Sinha N, Agrawal A, Pati AK. Role of ultrasound guided transversus abdominis plane block as a component of multimodal analgesic regimen for lower segment caesarean section: a randomized double blind clinical study. BMC Anesthesiol. 2018 May 14;18(1):53. doi: 10.1186/s12871-018-0512-x. PMID 29759061
- [Background] Aydin ME, Bedir Z, Yayik AM, Celik EC, Ates I, Ahiskalioglu EO, Ahiskalioglu A. Subarachnoid block and ultrasound-guided transversalis fascia plane block for caesarean section: A randomised, double-blind, placebo-controlled trial. Eur J Anaesthesiol. 2020 Sep;37(9):765-772. doi: 10.1097/EJA.0000000000001222. PMID 32412986
- [Derived] Pinarbasi A, Altiparmak B, Korkmaz Toker M, Pirincci F, Ugur B. Ultrasound-guided transversalis fascia plane block or transversus abdominis plane block for recovery after caesarean section: A randomised clinical trial. Eur J Anaesthesiol. 2024 Oct 1;41(10):769-778. doi: 10.1097/EJA.0000000000002041. Epub 2024 Jul 22. PMID 39039833